CLINICAL TRIAL: NCT07279727
Title: Ultrasound-Guided Infraclvicular Block Using Dexmedetomidine Versus Nalbuphine as Adjuvants to Bupivacaine in Upper Limb Orthopedic Surgery: A Prospective, Randomized, Double-Blind Controlled Study
Brief Title: Ultrasound-Guided Infraclvicular Block Using Dexmedetomidine Versus Nalbuphine as Adjuvants to Bupivacaine in Upper Limb Orthopedic Surgery
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mo'men mostafa youssef, Lecturer of Anesthesia and icu, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Infraclavicular nerve block
Record Dates: First submitted 2025-11-27; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Regional Anaesthesia
Keywords: Nalbuphine; Dexmedetomidine; Duration of analgesia; Bupivacaine; Infraclavicular block
MeSH Terms: interventions — Nalbuphine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nalbuphine group (Active Comparator): • Patients in group N (Nalbuphine group) will receive 29 mL of 0.5% bupivacaine + 1 mL (containing 10 mg nalbuphine)
  Interventions: Drug: Nalbuphine
- Dexmedetomidine group (Active Comparator): • Patients in group D (Dexmedetomidine group) will receive 29 mL of 0.5% bupivacaine + 1mL (containing 75 µg dexmedetomidine
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Nalbuphine — Nalbuphine will be added to .5% bupivacaine as an adjuvant in infraclavicular nerve block
  Arms: nalbuphine group
Drug: Dexmedetomidine — Dexmedetomidine will be added to .5% bupivacaine as an adjuvant in infraclavicular nerve block
  Other Names: precedex
  Arms: Dexmedetomidine group

SUMMARY:
this study is designed to evaluate and compare the efficacy of dexmedetomidine and nalbuphine as adjuvants to 0.5% bupivacaine in ultrasound-guided infraclavicular brachial plexus block for patients undergoing elective upper limb orthopedic surgeries on the duration of analgesia.

DETAILED DESCRIPTION:
Regional anesthesia is an integral component of modern anesthetic practice. It provides high-quality surgical anesthesia and superior postoperative analgesia while avoiding airway manipulation, minimizing systemic opioid use, and facilitating early ambulation and discharge .

Compared with general anesthesia, regional techniques reduce postoperative pain scores, nausea, and opioid requirements, leading to faster recovery and higher patient satisfaction. They are especially valuable in orthopedic upper-limb surgeries where prolonged postoperative analgesia is desired.

For upper limb procedures, various brachial plexus approaches-interscalene, supraclavicular, infraclavicular, and axillary-are utilized depending on the surgical site. Ultrasound guidance has greatly improved the safety and success rates of these blocks by allowing direct visualization of the nerves, needle, and spread of local anesthetic (LA).

The infraclavicular approach targets the cords of the brachial plexus surrounding the axillary artery in the infraclavicular fossa. It provides dense anesthesia and analgesia for surgeries of the elbow, forearm, and hand. Advantages over the supraclavicular or axillary approaches include reliable blockade of the musculocutaneous, median, ulnar, and radial nerves with a single injection, Lower risk of pneumothorax or phrenic nerve palsy and better catheter stability for continuous analgesia .

Despite these benefits, the main limitation is the finite duration of analgesia when using local anesthetics alone. Adjuvants have been explored to extend block duration and enhance quality without increasing toxicity. Commonly used agents include opioids, clonidine, dexmedetomidine, magnesium sulfate, dexamethasone, and others.

Dexmedetomidine is a highly selective α₂-adrenergic receptor agonist with sedative, anxiolytic, and analgesic properties and minimal respiratory depression.

It acts centrally through activation of α₂ receptors in the locus coeruleus inhibits norepinephrine release, producing sedation (Brummett et al., 2009) , and has peripheral action through hyperpolarization of C and Aδ nerve fibers via inhibition of sodium and potassium channels prolongs the effect of local anesthetics.

The addition of Dexmedetomidine as adjuvant to local bupivacaine in regional anesthesia has proven to : Shortens onset time of sensory and motor block, Prolongs block duration and postoperative analgesia by 3-6 hours, Reduces rescue analgesic consumption, and Provides mild sedation without respiratory depression.

However, potential adverse effects include bradycardia and hypotension related to systemic absorption, particularly at higher doses.

Nalbuphine hydrochloride is a synthetic opioid agonist-antagonist that acts predominantly as a κ-receptor agonist and µ-receptor antagonist. This pharmacologic profile provides potent analgesia with limited risk of respiratory depression, pruritus, or nausea commonly associated with pure µ-agonists such as morphine or fentanyl.

When used as an adjuvant to local anesthetics, nalbuphine is thought to: Prolong sensory and motor block duration, increase postoperative analgesia, Reduce opioid consumption, and has Minimal side effects . it produce its effects through acting on opioid receptors located on peripheral sensory nerve endings and by reducing inflammatory mediator release.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18-65 years ASA I-II (American Society of Anesthesiologists physical status classification) Scheduled for elective upper limb orthopedic surgeries Able to provide informed consent to participate in the study

Exclusion Criteria:

Refusal to participate in the study Pregnancy Allergy to any study drug(s) Neurological disease (e.g., neuropathies, central nervous system disorders) Coagulopathy or active bleeding disorders Severe systemic diseases (e.g., uncontrolled cardiovascular, renal, or liver disease) Opioid abuse or history of substance use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Our primary outcome of this study will be: Duration of Analgesia. | till 24 hour postoperative
  Definition: The time interval (in minutes) between the completion of the infraclavicular block injection and the first request for rescue analgesia (VAS ≥ 3).
  Scale: Visual Analog Scale (VAS)
  Scale Title: Visual Analog Scale for Pain (VAS)
  Minimum Value: 0 (no pain)
  Maximum Value: 10 (worst possible pain)
  Interpretation: Higher VAS scores indicate worse pain, and a score of ≥ 3 indicates the need for rescue analgesia.

SECONDARY OUTCOMES:
Onset time of sensory and motor block | till 20 minute after the block
Duration of sensory and motor block | 20 minute after the block
Time to first rescue analgesic request | till 24 hour postoperative
Heart rate (HR) | till 24 hour postoperative
Mean arterial blood pressure (MAP) | 24 hour postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Momen mostafa meki, Dr, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine Assiut University, Assiut,, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes